CLINICAL TRIAL: NCT03226678
Title: An Open Label, Prospective, Study to Assess the Safety, Tolerability, Efficacy and Pharmacokinetics of APL-2 in Patients With Warm Type Autoimmune Hemolytic Anemia (wAIHA) or Cold Agglutinin Disease (CAD)
Brief Title: Study to Assess the Safety, Tolerability, Efficacy and PK of APL-2 in Patients With Warm Type Autoimmune Hemolytic Anemia (wAIHA) or Cold Agglutinin Disease (CAD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Apellis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APL2-CP-AIHA-208
Record Dates: First submitted 2017-07-07; First posted 2017-07-24 (Actual); Results first posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-11

CONDITIONS: Warm Autoimmune Hemolytic Anemia; Cold Agglutinin Disease
MeSH Terms: conditions — Anemia, Hemolytic, Autoimmune

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 270mg or 360mg APL-2 administered subcutaneously daily (CAD) (Experimental)
  Interventions: Drug: APL-2
- 270mg or 360mg APL-2 administered subcutaneously daily (wAIHA) (Experimental)
  Interventions: Drug: APL-2

INTERVENTIONS:
Drug: APL-2 — Complement (C3) Inhibitor

SUMMARY:
This study is to assess the safety, tolerability, preliminary efficacy, and pharmacokinetics of APL-2 in subjects with warm Autoimmune Hemolytic Anemia (wAIHA) or Cold Agglutinin Disease (CAD).

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age.
2. Weight < 125 Kg.
3. Subjects must have a primary diagnosis of wAIHA or CAD defined by the presence of hemolytic anemia and positive DAT for wAIHA (IgG) or CAD (C3).
4. Hemoglobin <11 g/dL.
5. Signs of hemolysis with abnormal values by any of the hemolytic markers:

   1. Increased absolute reticulocyte count (above ULN)
   2. Reduced haptoglobin (below LLN)
   3. Increased lactase dehydrogenase (LDH) (above ULN)
   4. Increased indirect bilirubin (above ULN)
6. Women of child-bearing potential (WOCBP) (defined as any female who has experienced menarche and who is NOT permanently sterile or postmenopausal. Postmenopausal is defined as 12 consecutive months with no menses without an alternative medical cause) must have a negative pregnancy test at screening and must agree to use protocol defined methods of contraception for the duration of the study and 60 days after their last dose of study drug.
7. Males must agree to use protocol defined methods of contraception and agree to refrain from donating sperm for the duration of the study and 60 days after their last dose of study drug.
8. Able to provide documentary evidence of the following vaccinations within 2 years prior to screening:

   1. Neisseria meningitides types A, C, W, Y and type B (administered as two separate vaccinations)
   2. Streptococcus pneumoniae (Pneumococcal conjugate vaccine and Pneumococcal polysaccharide vaccine 23 [PCV13 and/or PPSV23, respectively])
   3. Haemophilus influenzae Type B (Hib) vaccine

   Subjects that do not have documentary evidence must be willing to receive any missing vaccinations as outlined below:
   1. Neisseria meningitides types A, C, W, Y and type B must be administered prior to dosing on Day 1. A booster is administered after at least 8 weeks (Day 56; for both vaccinations).
   2. Streptococcus pneumoniae PCV13 must be administered prior to dosing on Day 1 (see Section 12.2 for details). A PPSV23 booster is administered after at least 8 weeks (Day 56)
   3. Haemophilus influenze Type B (Hib) must be administered prior to dosing on Day 1.
9. Willing and able to give informed consent.
10. Specific for wAIHA: Relapsed from, did not respond or relapsed, or did not tolerate, at least one prior wAIHA treatment regimen (such as prednisone, rituximab).

Exclusion Criteria:

1. Prior treatment with rituximab within 90 days.
2. Deficiency of iron, folic acid and vitamin B12 prior to treatment phase
3. Abnormal liver function as indicated by a direct bilirubin above normal level, and/or an AST or ALT level > 2x upper limit of normal. Please note elevated indirect bilirubin due to hemolysis is not an exclusion criteria.
4. Elevated bilirubin not due to active hemolysis. Any elevation of bilirubin >ULN will require Sponsor review and approval for subject enrollment into the trial.
5. Active aggressive lymphoma requiring therapy or an active non-lymphatic malignant disease other than basal cell carcinoma or carcinoma in situ (CIS) of the cervix.
6. Presence or suspicion of active bacterial or viral infection, in the opinion of the Investigator, at screening or severe recurrent bacterial infections.
7. Participation in any other investigational drug trial or exposure to other investigational agent, device, or procedure within 30 days prior to screening period.
8. Pregnant, breast-feeding, or intending to conceive during the course of the study, including the Post-Treatment Phase.
9. Inability to cooperate or any condition that, in the opinion of the investigator, could increase the subject's risk by participating in the study or confound the outcome of the study.
10. Myocardial infarction, CABG, coronary or cerebral artery stenting and /or angioplasty, stroke, cardiac surgery, or hospitalization for congestive heart failure within 3 months or > Class 2 Angina Pectoris or NYHA Heart Failure Class >2
11. QTcF > 470 ms
12. PR > 280 ms
13. Mobitz II 2nd degree AV Block, 2:1 AV Block, High Grade AV Block, or Complete Heart Block unless the patient has an implanted pacemaker or implantable cardiac defibrillator (ICD) with backup pacing capabilities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-08-31 (Actual); Primary Completion 2022-09-12 (Actual); Study Completion 2022-09-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - American Institute of Research, Whittier, California
  - Lakes Research, Miami Lakes, Florida
  - Mid Florida Hematology Oncology, Orange City, Florida
  - University of Iowa Hospitals, Iowa City, Iowa
  - Mayo Clinic, Rochester, Minnesota
  - East Carolina University, Greenville, North Carolina
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Northwest Medical Specialties, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Roman E, Fattizzo B, Shum M, Hanna W, Lentz SR, Araujo SSS, Al-Adhami M, Grossi FV, Gertz MA. Safety and efficacy of pegcetacoplan treatment for cold agglutinin disease and warm antibody autoimmune hemolytic anemia. Blood. 2025 Jan 23;145(4):397-408. doi: 10.1182/blood.2023022549. PMID 39486046

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase 2, prospective pilot study was conducted at 12 sites in Brazil and United States of America in subjects with primary diagnosis of warm antibody autoimmune hemolytic anemia (wAIHA) or cold agglutinin disease (CAD) in parallel between 27 March 2018 and 12 September 2022.
Pre-assignment Details: The study consisted of 2 parts: Part A (core study phase; 12 months) and Part B (long-term extension phase; until the subject discontinued or the development program was terminated). Subjects were screened within 30 days prior to the start of dosing on day 1. A total of 24 subjects were enrolled.
Groups:
- Part A: Cohort 1 wAIHA - 270 mg: Subjects diagnosed with wAIHA received pegcetacoplan 270 milligram (mg) per day subcutaneous (SC) infusion up to 12 months in Part A.
- Part A: Cohort 1 wAIHA - 360 mg: Subjects diagnosed with wAIHA received pegcetacoplan 360 mg per day SC infusion up to 12 months in Part A.
- Part A: Cohort 2 CAD - 270 mg: Subjects diagnosed with CAD received pegcetacoplan 270 per day SC infusion up to 12 months in Part A.
- Part A: Cohort 2 CAD - 360 mg: Subjects diagnosed with CAD received pegcetacoplan 360 mg per day SC infusion up to 12 months in Part A.
- Part B: Cohort 1 wAIHA - 1080 mg: Eligible subjects diagnosed with wAIHA from Part A entered Part B to receive pegcetacoplan 1080 mg SC infusion twice weekly (with the potential to escalate to 1080 mg every 3 days) until the subject discontinued or the development program was terminated.
- Part B: Cohort 2 CAD - 1080 mg: Eligible subjects diagnosed with CAD from Part A entered Part B to receive pegcetacoplan 1080 mg SC infusion twice weekly (with the potential to escalate to 1080 mg every 3 days) until the subject discontinued or the development program was terminated.
Period: Part A (Core Study Phase)
Arm/Group | Part A: Cohort 1 wAIHA - 270 mg | Part A: Cohort 1 wAIHA - 360 mg | Part A: Cohort 2 CAD - 270 mg | Part A: Cohort 2 CAD - 360 mg | Part B: Cohort 1 wAIHA - 1080 mg | Part B: Cohort 2 CAD - 1080 mg
Started | 5 | 6 | 7 | 6 | 0 | 0
Completed | 3 | 3 | 5 | 5 | 0 | 0
Not Completed | 2 | 3 | 2 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Non-compliance with study drug | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrew, per Investigator | 2 | 1 | 0 | 0 | 0 | 0
Period: Part B (Long-Term Extension Phase)
Arm/Group | Part A: Cohort 1 wAIHA - 270 mg | Part A: Cohort 1 wAIHA - 360 mg | Part A: Cohort 2 CAD - 270 mg | Part A: Cohort 2 CAD - 360 mg | Part B: Cohort 1 wAIHA - 1080 mg | Part B: Cohort 2 CAD - 1080 mg
Started | 0 (Eligible subjects entered Part B.) | 0 (Eligible subjects entered Part B.) | 0 (Eligible subjects entered Part B.) | 0 (Eligible subjects entered Part B.) | 5 (Eligible subjects from 'Part A: Cohort 1 wAIHA - 270 mg' and 'Part A: Cohort 1 wAIHA - 360 mg' reporting groups entered Part B.) | 9 (Eligible subjects from 'Part A: Cohort 2 CAD - 270 mg' and 'Part A: Cohort 2 CAD - 360 mg' reporting groups entered Part B.)
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 5 | 9
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 2 | 1
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Non-Compliance With Study Drug | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Study Terminated By Sponsor | 0 | 0 | 0 | 0 | 3 | 5
Not completed — Withdrew, Per Sponsor | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Safety set included all subjects who received at least 1 dose of study drug.
Groups:
- Part A: Cohort 1 wAIHA - 270 mg: Subjects diagnosed with wAIHA received pegcetacoplan 270 mg per day SC infusion up to 12 months in Part A.
- Total: Total of all reporting groups
Arm/Group | Part A: Cohort 1 wAIHA - 270 mg | Part A: Cohort 1 wAIHA - 360 mg | Part A: Cohort 2 CAD - 270 mg | Part A: Cohort 2 CAD - 360 mg | Total
Number analyzed (Participants) | 5 | 6 | 7 | 6 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.6 (17.57) | 54.3 (22.12) | 68.9 (8.51) | 75.7 (7.53) | 64.8 (16.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 4 | 5 | 15
  Male | 2 | 3 | 3 | 1 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black Or African American | 0 | 0 | 0 | 1 | 1
  White | 5 | 6 | 7 | 5 | 23
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic Or Latino | 3 | 3 | 1 | 1 | 8
  Not Hispanic Or Latino | 2 | 3 | 6 | 5 | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Treatment Emergent Adverse Events (TEAEs) Including by Severity
Description: TEAEs were defined as adverse events (AEs) that occurred after dosing on Day 1 and up to 56 days after the last dose of study drug. A treatment-related TEAE is defined as a TEAE with a relationship to study drug of probably, possibly, unlikely, or unrelated. A serious adverse event (SAE) is defined as any AE that resulted in death; was life-threatening; required hospitalization or prolongation of existing hospitalization; resulted in persistent or significant incapacity or substantial disruption of ability to conduct normal life functions; was a congenital anomaly or birth defect. TEAEs were graded according to Common Terminology Criteria for Adverse Events v4.03 based on: Grade 1: Mild; Grade 2: Moderate; Grade 3: Severe; Grade 4: Life-threatening; Grade 5: Death related to AE.
Time Frame: Part A:From first dose of study drug (Part A Day 1) up to 30days after last dose of study drug in Part A,approximately 366days Part B:From first dose of study drug (Part B Day 1) up to 56days after last dose of study drug in Part B,approximately 980days
Population: The Safety set included all subjects who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Cohort 1 wAIHA - 270 mg | Part A: Cohort 1 wAIHA - 360 mg | Part A: Cohort 2 CAD - 270 mg | Part A: Cohort 2 CAD - 360 mg | Part B: Cohort 1 wAIHA - 1080 mg | Part B: Cohort 2 CAD - 1080 mg
Number analyzed (Participants) | 5 | 6 | 7 | 6 | 5 | 9
Participants
  All TEAEs | 5 | 5 | 7 | 6 | 5 | 9
  Treatment related TEAEs | 4 | 4 | 5 | 4 | 4 | 5
  Serious AEs | 3 | 2 | 3 | 2 | 2 | 6
  TEAEs leading to study drug discontinuation | 1 | 2 | 1 | 1 | 2 | 2
  TEAEs leading to death | 0 | 0 | 1 | 0 | 0 | 1
  TEAEs with mild intensity | 2 | 1 | 0 | 0 | 1 | 1
  TEAEs with moderate intensity | 0 | 2 | 3 | 3 | 3 | 2
  TEAEs with severe intensity | 3 | 2 | 3 | 2 | 1 | 4
  TEAEs with life threatening intensity | 0 | 0 | 0 | 1 | 0 | 1

2. Secondary Outcome: Mean Change From Baseline in Hemoglobin at Weeks 48 and 132
Description: Hematology assessments of hemoglobin were made at the last measurement prior to the first dose of pegcetacoplan (baseline) and periodically throughout the different parts of the treatment period. Mean change from baseline in hemoglobin results were summarized from Part A baseline for Part A reporting groups and from Part B baseline for Part B reporting groups.
Time Frame: Part A: Baseline (Day 1 of Part A) and Week 48; Part B: Baseline (Day 1 of Part B) and Week 132
Population: The intent-to-treat (ITT) analysis set included all subjects who received at least 1 dose of study drug. Only subjects analyzed at specific timepoint are reported.
Measure: Mean (Standard Deviation); unit: gram per deciliter (g/dL)
Arm/Group | Part A: Cohort 1 wAIHA - 270 mg | Part A: Cohort 1 wAIHA - 360 mg | Part A: Cohort 2 CAD - 270 mg | Part A: Cohort 2 CAD - 360 mg | Part B: Cohort 1 wAIHA - 1080 mg | Part B: Cohort 2 CAD - 1080 mg
Number analyzed (Participants) | 4 | 3 | 6 | 4 | 2 | 4
gram per deciliter (g/dL)
  Week 48: number analyzed (Participants) | 4 | 3 | 6 | 4 | 0 | 0
  Week 48 | 0.38 (2.347) | 1.93 (0.874) | 1.62 (1.522) | 2.63 (1.694) |  |
  Week 132: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 4
  Week 132 |  |  |  |  | 0.18 (0.626) | -0.20 (2.029)

3. Secondary Outcome: Number of Subjects Who Received Red Blood Cell (RBC) Transfusions
Description: The number of on-study RBC transfusions were monitored throughout the treatment period.
Time Frame: From Day 1 up to Week 132
Population: The ITT analysis set included all subjects who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Cohort 1 wAIHA - 270 mg | Part A: Cohort 1 wAIHA - 360 mg | Part A: Cohort 2 CAD - 270 mg | Part A: Cohort 2 CAD - 360 mg | Part B: Cohort 1 wAIHA - 1080 mg | Part B: Cohort 2 CAD - 1080 mg
Number analyzed (Participants) | 5 | 6 | 7 | 6 | 5 | 9
Participants | 2 | 2 | 2 | 1 | 0 | 3

4. Secondary Outcome: Mean Change From Baseline in Absolute Reticulocyte Count (ARC) at Weeks 48 and 132
Description: Hematology assessments of ARC were made at the last measurement prior to the first dose of pegcetacoplan (baseline) and periodically throughout the different parts of the treatment period. Mean change from baseline in ARC results were summarized from Part A baseline for Part A reporting groups and from Part B baseline for Part B reporting groups.
Time Frame: Part A: Baseline (Day 1 of Part A) and Week 48; Part B: Baseline (Day 1 of Part B) and Week 132
Population: The ITT analysis set included all subjects who received at least 1 dose of study drug. Only subjects analyzed at specific timepoint are reported.
Measure: Mean (Standard Deviation); unit: 10^9 cells/liter (L)
Arm/Group | Part A: Cohort 1 wAIHA - 270 mg | Part A: Cohort 1 wAIHA - 360 mg | Part A: Cohort 2 CAD - 270 mg | Part A: Cohort 2 CAD - 360 mg | Part B: Cohort 1 wAIHA - 1080 mg | Part B: Cohort 2 CAD - 1080 mg
Number analyzed (Participants) | 4 | 3 | 4 | 5 | 2 | 4
10^9 cells/liter (L)
  Week 48: number analyzed (Participants) | 4 | 3 | 4 | 5 | 0 | 0
  Week 48 | -145.050 (90.4181) | -130.187 (70.4638) | -73.515 (73.1983) | -84.064 (46.0655) |  |
  Week 132: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 4
  Week 132 |  |  |  |  | 11.485 (4.9787) | 81.585 (83.4790)

5. Secondary Outcome: Mean Change From Baseline in Lactate Dehydrogenase (LDH) at Weeks 48 and 132
Description: Serum chemistry assessments of LDH were made at the last measurement prior to the first dose of pegcetacoplan (baseline) and periodically throughout the different parts of the treatment period. Mean change from baseline in LDH results were summarized from Part A baseline for Part A reporting groups and from Part B baseline for Part B reporting groups.
Time Frame: Part A: Baseline (Day 1 of Part A) and Week 48; Part B: Baseline (Day 1 of Part B) and Week 132
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: international units/L
Arm/Group | Part A: Cohort 1 wAIHA - 270 mg | Part A: Cohort 1 wAIHA - 360 mg | Part A: Cohort 2 CAD - 270 mg | Part A: Cohort 2 CAD - 360 mg | Part B: Cohort 1 wAIHA - 1080 mg | Part B: Cohort 2 CAD - 1080 mg
Number analyzed (Participants) | 4 | 3 | 5 | 5 | 2 | 4
international units/L
  Week 48: number analyzed (Participants) | 4 | 3 | 5 | 5 | 0 | 0
  Week 48 | -51.8 (39.08) | -169.7 (212.89) | -475.8 (842.43) | -77.8 (73.30) |  |
  Week 132: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 4
  Week 132 |  |  |  |  | 1.78 (46.357) | 35.18 (82.727)

6. Secondary Outcome: Mean Change From Baseline in Haptoglobin at Weeks 48 and 132
Description: Serum chemistry assessments of haptoglobin were made at the last measurement prior to the first dose of pegcetacoplan (baseline) and periodically throughout the different parts of the treatment period. Mean change from baseline in haptoglobin results were summarized from Part A baseline for Part A reporting groups and from Part B baseline for Part B reporting groups.
Time Frame: Part A: Baseline (Day 1 of Part A) and Week 48; Part B: Baseline (Day 1 of Part B) and Week 132
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Part A: Cohort 1 wAIHA - 270 mg | Part A: Cohort 1 wAIHA - 360 mg | Part A: Cohort 2 CAD - 270 mg | Part A: Cohort 2 CAD - 360 mg | Part B: Cohort 1 wAIHA - 1080 mg | Part B: Cohort 2 CAD - 1080 mg
Number analyzed (Participants) | 4 | 3 | 6 | 5 | 2 | 4
g/L
  Week 48: number analyzed (Participants) | 4 | 3 | 6 | 5 | 0 | 0
  Week 48 | 0.715 (0.7622) | 0.747 (0.7306) | 0.528 (0.4961) | 0.172 (0.3404) |  |
  Week 132: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 4
  Week 132 |  |  |  |  | -0.270 (0.6364) | -0.335 (0.1323)

7. Secondary Outcome: Mean Change From Baseline in Indirect Bilirubin at Weeks 48 and 132
Description: Serum chemistry assessments of indirect bilirubin were made at the last measurement prior to the first dose of pegcetacoplan (baseline) and periodically throughout the different parts of the treatment period. Mean change from baseline in indirect bilirubin results were summarized from Part A baseline for Part A reporting groups and from Part B baseline for Part B reporting groups.
Time Frame: Part A: Baseline (Day 1 of Part A) and Week 48; Part B: Baseline (Day 1 of Part B) and Week 132
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: micromole/L
Arm/Group | Part A: Cohort 1 wAIHA - 270 mg | Part A: Cohort 1 wAIHA - 360 mg | Part A: Cohort 2 CAD - 270 mg | Part A: Cohort 2 CAD - 360 mg | Part B: Cohort 1 wAIHA - 1080 mg | Part B: Cohort 2 CAD - 1080 mg
Number analyzed (Participants) | 4 | 3 | 5 | 5 | 2 | 4
micromole/L
  Week 48: number analyzed (Participants) | 4 | 3 | 5 | 5 | 0 | 0
  Week 48 | -10.723 (4.2167) | -9.697 (5.2220) | -15.879 (15.1038) | -17.981 (7.0978) |  |
  Week 132: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 4
  Week 132 |  |  |  |  | 0.195 (0.2764) | 4.095 (8.7678)

8. Secondary Outcome: Maximum Observed Trough Serum Concentration (Ctrough,Max) of Pegcetacoplan
Description: Blood samples were collected for the assessment of Ctrough,max of pegcetacoplan.
Time Frame: Pre-dose and 4 hours postdose on Day 1; pre-dose on Weeks 1, 2, 4, 8, 12, 16, 20, 24, 32, 36, 40, 48, 60, 72, 84, 96, 108, 120 and 132
Population: The Pharmacokinetic analysis set included all subjects in the Safety set who had at least 1 evaluable post-dose pharmacokinetic measurement that was not below the limit of quantification.
Measure: Mean (Standard Deviation); unit: microgram per milliliter
Arm/Group | Part A: Cohort 1 wAIHA - 270 mg | Part A: Cohort 1 wAIHA - 360 mg | Part A: Cohort 2 CAD - 270 mg | Part A: Cohort 2 CAD - 360 mg | Part B: Cohort 1 wAIHA - 1080 mg | Part B: Cohort 2 CAD - 1080 mg
Number analyzed (Participants) | 5 | 6 | 7 | 6 | 5 | 9
microgram per milliliter | 629.6 (206.66) | 679.7 (303.76) | 661.6 (192.24) | 807.8 (105.12) | 813.6 (260.08) | 795.6 (204.90)

9. Secondary Outcome: Mean Change From Baseline in Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Score at Weeks 48 and 132
Description: The FACIT-Fatigue Scale is a 13 item Likert scaled instrument where the subject was presented with 13 statements and asked to indicate their response as it applied to the past 7 days. The 5 possible responses were 'Not at all' (0), 'A little bit (1), 'Somewhat' (2), 'Quite a bit' (3) and 'Very much' (4). There are 13 statements with the total score ranging from 0 to 52 and higher scores indicating better quality of life. Mean change from baseline in FACIT-Fatigue score results were summarized from Part A baseline for Part A reporting groups and from Part B baseline for Part B reporting groups.
Time Frame: Part A: Baseline (Day 1 of Part A) and Week 48; Part B: Baseline (Day 1 of Part B) and Week 132
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part A: Cohort 1 wAIHA - 270 mg | Part A: Cohort 1 wAIHA - 360 mg | Part A: Cohort 2 CAD - 270 mg | Part A: Cohort 2 CAD - 360 mg | Part B: Cohort 1 wAIHA - 1080 mg | Part B: Cohort 2 CAD - 1080 mg
Number analyzed (Participants) | 4 | 3 | 6 | 4 | 2 | 4
score on a scale
  Week 48: number analyzed (Participants) | 4 | 3 | 6 | 4 | 0 | 0
  Week 48 | -3.8 (8.38) | 10.7 (5.51) | 0.5 (16.33) | 9.0 (7.07) |  |
  Week 132: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 4
  Week 132 |  |  |  |  | -1.0 (1.41) | 2.8 (7.23)

10. Secondary Outcome: Mean Change From Baseline in Linear Analog Scale Assessment (LASA) Score at Weeks 48 and 132
Description: The LASA consists of 5 single statements asking subjects to rate their perceived level of functioning. Specific domains include physical well-being (fatigue, activity level), emotional well-being (depression, anxiety, stress), spiritual well-being (sense of meaning), and intellectual well-being (ability to think clearly and concentrate). An item for overall quality of life is also included. Each domain scale range from 0 to 10. Where, 0 = as bad as it can be and 10 = as good as it can be. The total score ranging from 0 to 50 and higher scores indicating better quality of life. Mean change from baseline in LASA score results were summarized from Part A baseline for Part A reporting groups and from Part B baseline for Part B reporting groups.
Time Frame: Part A: Baseline (Day 1 of Part A) and Week 48; Part B: Baseline (Day 1 of Part B) and Week 132
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part A: Cohort 1 wAIHA - 270 mg | Part A: Cohort 1 wAIHA - 360 mg | Part A: Cohort 2 CAD - 270 mg | Part A: Cohort 2 CAD - 360 mg | Part B: Cohort 1 wAIHA - 1080 mg | Part B: Cohort 2 CAD - 1080 mg
Number analyzed (Participants) | 4 | 3 | 6 | 4 | 2 | 4
score on a scale
  Week 48: number analyzed (Participants) | 4 | 3 | 6 | 4 | 0 | 0
  Week 48 | 0.0 (2.45) | 1.3 (4.04) | 0.8 (1.72) | 1.0 (1.15) |  |
  Week 132: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 4
  Week 132 |  |  |  |  | 0.0 (0.00) | 0.5 (1.73)

ADVERSE EVENTS:
Time Frame: Part A: TEAE data is reported from first dose of study drug (Day 1 of Part A) up to 30 days after the last dose of study drug in Part A, approximately 366 days. Part B: TEAE data is reported from first dose of study drug (Day 1 of Part B) up to 56 days after the last dose of study drug in Part B, approximately 980 days. All-cause mortality: From first dose of study drug (Day 1) up to end of the study, approximately 1346 days.
Description: The Safety set included all subjects who received at least 1 dose of study drug. MedDRA version for Part A was 20.0 and Part B was 23.0.
Arm/Group | Part A: Cohort 1 wAIHA - 270 mg | Part A: Cohort 1 wAIHA - 360 mg | Part A: Cohort 2 CAD - 270 mg | Part A: Cohort 2 CAD - 360 mg | Part B: Cohort 1 wAIHA - 1080 mg | Part B: Cohort 2 CAD - 1080 mg
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/6 | 1/7 | 0/6 | 0/5 | 1/9
Serious Adverse Events (participants affected / at risk) | 3/5 | 2/6 | 3/7 | 2/6 | 2/5 | 6/9
Other Adverse Events (participants affected / at risk) | 5/5 | 5/6 | 7/7 | 6/6 | 5/5 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Cohort 1 wAIHA - 270 mg (N=5) | Part A: Cohort 1 wAIHA - 360 mg (N=6) | Part A: Cohort 2 CAD - 270 mg (N=7) | Part A: Cohort 2 CAD - 360 mg (N=6) | Part B: Cohort 1 wAIHA - 1080 mg (N=5) | Part B: Cohort 2 CAD - 1080 mg (N=9)
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 2 | 0 | 1 | 0 | 0 | 0
Haemolysis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Gastritis erosive (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Blood calcium increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Generalised anxiety disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hip arthroplasty (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Cohort 1 wAIHA - 270 mg (N=5) | Part A: Cohort 1 wAIHA - 360 mg (N=6) | Part A: Cohort 2 CAD - 270 mg (N=7) | Part A: Cohort 2 CAD - 360 mg (N=6) | Part B: Cohort 1 wAIHA - 1080 mg (N=5) | Part B: Cohort 2 CAD - 1080 mg (N=9)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0 | 1 | 2
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2 | 0
Extravascular haemolysis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cyanosis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cerumen impaction (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0
Excessive cerumen production (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0
Goitre (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0
Thyroid mass (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 1 | 0 | 0 | 1 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Eye irritation (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Ocular hypertension (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 2 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 4 | 1 | 2 | 0
Diverticulum (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Gastric polyps (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 2 | 2 | 2 | 1
Oesophageal motility disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 1 | 1 | 2 | 1 | 1 | 2
Infusion site pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Infusion site rash (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Injection site bruising (General disorders) | 0 | 1 | 1 | 1 | 1 | 0
Injection site erythema (General disorders) | 1 | 1 | 1 | 1 | 1 | 1
Injection site pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Injection site pruritus (General disorders) | 2 | 1 | 0 | 1 | 0 | 1
Injection site reaction (General disorders) | 0 | 1 | 0 | 1 | 0 | 1
Injection site swelling (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Local swelling (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Oedema (General disorders) | 0 | 0 | 1 | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0 | 1 | 0
Pain (General disorders) | 1 | 1 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 2 | 2 | 1 | 1 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 1 | 0
Seasonal allergy (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Ear infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Incision site abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Mastitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Oral fungal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 2 | 3
Viral upper respiratory tract infection (Infections and infestations) | 1 | 1 | 1 | 2 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 3 | 1 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 1 | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Pseudophakic bullous keratopathy (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 2
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Blood cholesterol increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Blood glucose abnormal (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Blood phosphorus decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 4
White blood cell count decreased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Folate deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 1
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vitamin B complex deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 | 1 | 3 | 1 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 2 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Sinonasal papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 3 | 0 | 3
Headache (Nervous system disorders) | 0 | 0 | 3 | 1 | 3 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 1
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 2 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Generalised anxiety disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 1
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 0 | 1
Chromaturia (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Renal cyst (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Renal injury (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Renal mass (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Breast fibrosis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Uterine haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 2 | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 1 | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0
Lichenoid keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Skin warm (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Venous ulcer pain (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Flushing (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 1 | 3 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Leriche syndrome (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pallor (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Raynaud's phenomenon (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Spider vein (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-01-17): https://cdn.clinicaltrials.gov/large-docs/78/NCT03226678/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-27): https://cdn.clinicaltrials.gov/large-docs/78/NCT03226678/SAP_001.pdf